CLINICAL TRIAL: NCT02373943
Title: Bioavailability of Vitamin A From β-carotene-Biofortified Maize Porridge Consumed by Women and Men: Results of a Randomized Crossover Trial
Brief Title: The MULTINUTRIENT Maize Project: Results of Human Feeding Trial
Acronym: MAIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Joan Antoni Schoenenberger, Dr. Joan Antoni Schoenenberger Arnaiz, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ERCEA - PoC2013 - 619161
Record Dates: First submitted 2015-02-15; First posted 2015-02-27 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: vitamin A; human; bioavailability; fortified maize; cross-over; beta-carotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- β-carotene biofortified maize (Experimental): Participants will ingest porridge bF: this will be the β-carotene fortified maize porridge where each 250 g will be made with 50 g of dry maize flour obtained from fortified corn seeds. The contents of β-carotene and other provitamin A carotenoids in this flour will be determined before preparing the porridges.
  Interventions: Other: β-carotene biofortified maize
- white maize supplemented with β-carotene (Active Comparator): Participants will ingest porridge F: this will be also a β-carotene fortified maize porridge but in this case it will be made with 50 g of dry maize flour obtained from non fortified corn seeds and supplemented with a 500-1500 µg β-carotene reference dose. The exact dose of β-carotene that will be added to these porridges will be established according to the amount of β-carotene found in the flour used with porridges BF.
  Interventions: Other: β-carotene supplemented maize
- white maize (Sham Comparator): Participants will ingest porridge N which will be the control porridge and will be made with 50 g of dry maize flour obtained from non fortified corn seeds.
  Interventions: Other: Normal (non biofortified) maize without added β-carotene

INTERVENTIONS:
Other: β-carotene biofortified maize — Determination of all-trans retinol AUC values after the ingestion of 200 g porridge made with 50 g of flour of β-carotene fortified maize
  Arms: β-carotene biofortified maize
Other: β-carotene supplemented maize — Determination of all-trans retinol AUC values after the ingestion of 200 g porridge made with 50 g of flour of β-carotene supplemented maize
  Arms: white maize supplemented with β-carotene
Other: Normal (non biofortified) maize without added β-carotene — Determination of all-trans retinol AUC values after the ingestion of 200 g porridge made with 50 g of flour of normal maize
  Arms: white maize

SUMMARY:
The main objective of this human trial is the demonstration that β-carotene in fortified maize has good bioavailability as a plant source of vitamin A and that when humans ingest the biofortified product retinol levels are higher than when they ingest non biofortified white maize.

DETAILED DESCRIPTION:
Human feeding trial with fortified maize is part of the BIOFORCE project which aims to create transgenic cereal plants that will provide a near complete micronutrient complement for malnourished people. β-Carotene intake helps to balance inadequate retinol supply in significant parts of the world. In order for plants with enhanced levels of micronutrients to be useful, the micronutrients must be present in a bioavailable form that can be absorbed by the human body. To test the main hypothesis of the trial an open-label, randomized, three-way crossover trial consisting of three 7-day feeding periods has been designed. The study will compare three different feeding conditions: β-carotene fortified maize containing diet, white maize containing diet supplemented with a reference β-carotene dose and white maize diet. The study will test the hypothesis that a meal including fortified maize yields superior all-trans retinol area under the plasma concentration versus time curve (AUC) values than an isocaloric and isoprotein meal with normal maize.

After a first screen that will address physical conditions and lifestyle 18 volunteers (9 men and 9 women) who meet the eligibility criteria will be included in the study once they have read and sign the informed consent. The postprandial plasma all-trans retinol response to each test meal will be used to establish the bioavailability of provitamin A from fortified maize. The test meals will be consumed in random order separated by 1 week. Blood samples will be collected over 8 h. All-trans retinol will be analyzed in plasma by high pressure liquid chromatography (HPLC) with coulometric array electrochemical detection.

Mean AUC for all-trans retinol in plasma after ingestion of the β-carotene-fortified maize porridge, the white maize porridge with the β-carotene reference dose, and the white maize porridge will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons
* Persons who had not taken vitamin A or β-carotene supplements within the past month

Exclusion Criteria:

* Current or recent (previous 12 mo) cigarette smoking
* Frequent consumption of alcoholic beverages (1 drink/d)
* Current or recent (previous 1 mo) use of dietary supplements
* Current or recent (previous 6 mo) use of hormonal contraceptives
* Current or recent (previous 1 mo) use of medications known to affect lipid metabolism.
* History of restrictive eating
* BMI under 20 or over 30
* Lactose intolerance
* Vegetarians.
* Severe or symptomatic cardiac disease or hypertension
* History of bleeding disorders
* Chronic history of gastric, intestinal, liver, pancreatic, or renal disease
* Any portion of the stomach or the intestine removed (other than an appendectomy)
* History of intestinal obstruction, malabsorption, or use of antacid drugs; cancer (active or use of medications for a history of cancer treatment within the past 5 y)
* History of chronic alcoholism
* History of convulsive disorder
* Evidence of active drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of vitamin A bioavailability, as measured by the plasma all-trans retinol response, between fortified maize and wild type | Pharmacokinetic measures: -15 min, 2h, 3.5h, 5h, 7h. 8h
  Comparison of baseline corrected AUC plasma concentrations of all-trans retinol over 8h

SECONDARY OUTCOMES:
Relative bioavailability of provitamin A in terms of fortified maize vs wild type maize supplemented with a beta-carotene reference dose. | Pharmacokinetic measures: -15 min, 2h, 3.5h, 5h, 7h. 8h
  Comparison of baseline corrected AUC plasma concentrations of all-trans retinol over 8h

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Schoenenberger, Pharm D, Principal Investigator — Institut de Recerca Biomèdica de Lleida
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, LLeida, Spain

REFERENCES:
- [Background] Li S, Nugroho A, Rocheford T, White WS. Vitamin A equivalence of the ss-carotene in ss-carotene-biofortified maize porridge consumed by women. Am J Clin Nutr. 2010 Nov;92(5):1105-12. doi: 10.3945/ajcn.2010.29802. Epub 2010 Sep 1. PMID 20810977
- [Background] Grune T, Lietz G, Palou A, Ross AC, Stahl W, Tang G, Thurnham D, Yin SA, Biesalski HK. Beta-carotene is an important vitamin A source for humans. J Nutr. 2010 Dec;140(12):2268S-2285S. doi: 10.3945/jn.109.119024. Epub 2010 Oct 27. PMID 20980645
- [Background] Christou P, Twyman RM. The potential of genetically enhanced plants to address food insecurity. Nutr Res Rev. 2004 Jun;17(1):23-42. doi: 10.1079/NRR200373. PMID 19079913
- [Background] Paine JA, Shipton CA, Chaggar S, Howells RM, Kennedy MJ, Vernon G, Wright SY, Hinchliffe E, Adams JL, Silverstone AL, Drake R. Improving the nutritional value of Golden Rice through increased pro-vitamin A content. Nat Biotechnol. 2005 Apr;23(4):482-7. doi: 10.1038/nbt1082. Epub 2005 Mar 27. PMID 15793573
- [Background] Gannon B, Kaliwile C, Arscott SA, Schmaelzle S, Chileshe J, Kalungwana N, Mosonda M, Pixley K, Masi C, Tanumihardjo SA. Biofortified orange maize is as efficacious as a vitamin A supplement in Zambian children even in the presence of high liver reserves of vitamin A: a community-based, randomized placebo-controlled trial. Am J Clin Nutr. 2014 Dec;100(6):1541-50. doi: 10.3945/ajcn.114.087379. Epub 2014 Oct 8. PMID 25411289